CLINICAL TRIAL: NCT06489600
Title: Open-Label, Interventional, Prospective, Safety, In-Use Tolerability Study of Test Product "No Rays, Thanks Mineral Sunscreen" in Healthy Adult Subjects With Dry and Sensitive Skin.
Brief Title: A Clinical Study to Assess the Safety, In-use Tolerability of Test Product in Healthy Adult Subjects With Dry and Sensitive Skin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Kayura Effects LLP (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB240031-KE
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dry Skin; Sensitive Skin

STUDY DESIGN:
Intervention Model Description: open-label, interventional, prospective, safety in-use tolerability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No Rays, Thanks Mineral sunscreen (Experimental): Wash your face with standard facewash and apply a pea size amount on the face in the morning.
  Interventions: Other: No Rays, Thanks Mineral sunscreen

INTERVENTIONS:
Other: No Rays, Thanks Mineral sunscreen — Wash your face with standard facewash and apply a pea size amount on the face in the morning.
  Dosage form: semi-solid frequency: Once in a day Route of Administration: Topical

SUMMARY:
This is open-label, interventional, prospective, safety in-use tolerability study of test product "No Rays, Thanks Mineral Sunscreen" in healthy adult human subjects with dry and sensitive skin.

DETAILED DESCRIPTION:
A total of 27 subjects with preferably equal number of males and non-pregnant /non-lactating females will be enrolled to ensure a total of 25 subjects complete the study.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called on the telephone by the recruiting department prior to the enrolment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up on the study visit day. The adult male and female subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Day 01): Screening, Enrolment, Baseline Evaluation, on site product usage, Post usage evaluation at T15 mins.
* Visit 02 (Day 15 ±2 Days): Evaluations, End of Study

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 55 years (both inclusive) at the time of consent.
2. Sex: Healthy male and non-pregnant/non-lactating females. (Preferably equal ratio of males and females)
3. Females of childbearing potential must have a self-reported negative pregnancy test.
4. Subject are generally in good health.
5. Subject with dry and sensitive skins. (As per the dermatological evaluation).
6. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
7. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
8. Subjects are willing to give written informed consent and are willing to come for regular follow up.
9. Subjects who commit not to use medicated skincare products other than the test product for the entire duration of the study.
10. Subject who have not participated in a similar investigation in the past three months.
11. Willing to use test product throughout the study period.

Exclusion Criteria:

1. History of any dermatological condition of the skin disease.
2. Subject with present condition of allergic response to any cosmetic product.
3. Subjects under chronic medication (e.g. aspirin-based products, anti-inflammatories, anti-histamines, corticotherapy etc.) that might influence the outcome of the study.
4. History of alcohol or drug addiction.
5. The subject has clinically significant skin disease, which may contraindicate participation, including psoriasis, eczema, skin cancer or other skin pathology.
6. Subjects having skin infections like bacterial, fungal, viral infections.
7. The subject has skin irritation, open wounds, cuts, abrasions, irritation symptoms or any dermatological condition on the face that can interfere with the reading.
8. Be wearing any facial makeup, including false eyelashes, on the day of the study visit.
9. Subjects having hypersensitive skin.
10. Subjects using other marketed sun screen products during the study period.
11. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
12. Pregnant or breastfeeding or planning to become pregnant during the study period.
13. History of chronic illness which may influence the cutaneous state.
14. Subjects participating in other similar cosmetics, devices or therapeutic trials or skincare products within the last four weeks.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Change in local intolerance assessment for skin irritation using 4-point scoring scale where 0 indicate absent and 3 indicate severe. | On Day 01 at T15 minutes and on Day 15 (± 2 Days).
  To assess the safety of the test product in terms of change in local intolerance assessment for irritation by dermatological assessment
Change in local intolerance assessment for skin dryness using 4-point scoring scale where 0 indicate absent and 3 indicate severe. | On Day 01 at T15 minutes and on Day 15 (± 2 Days).
  To assess the safety of the test product in terms of change in local intolerance assessment for dryness by dermatological assessment
Change in local intolerance assessment for skin oedema using 4-point scoring scale where 0 indicate absent and 3 indicate severe. | On Day 01 at T15 minutes and on Day 15 (± 2 Days).
  To assess the safety of the test product in terms of change in local intolerance assessment for oedema by dermatological assessment
safety of the test product in terms of local intolerance assessment of irritation (Patient Global Assessment scale) where 0 indicate not at all and 10 indicate very severe. | On Day 01 at T15 minutes and on Day 15 (± 2 Days).
  To evaluate the safety of the test product in terms of local intolerance assessment of irritation by Patient Global Assessment scale.
safety of the test product in terms of local intolerance assessment of dryness (Patient Global Assessment scale) where 0 indicate not at all and 10 indicate very severe. | On Day 01 at T15 minutes and on Day 15 (± 2 Days).
  To evaluate the safety of the test product in terms of local intolerance assessment of dryness by Patient Global Assessment scale.
safety of the test product in terms of local intolerance assessment of oedema (Patient Global Assessment scale) where 0 indicate not at all and 10 indicate very severe. | On Day 01 at T15 minutes and on Day 15 (± 2 Days).
  To evaluate the safety of the test product in terms of local intolerance assessment of oedema by Patient Global Assessment scale.

SECONDARY OUTCOMES:
where will you rank the test product in terms of appearance in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters- appearance through the subject product perception assessment.
where will you rank the test product in terms of spreadibility in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters- spreadibility through the subject product perception assessment.
where will you rank the test product in terms of texture in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters-texture through the subject product perception assessment.
where will you rank the test product in terms of fragrance in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters-fragrance through the subject product perception assessment.
where will you rank the test product in terms of absorption in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters-absorption through the subject product perception assessment.
where will you rank the test product in terms of colour in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters-colour, through the subject product perception assessment.
where will you rank the test product in terms of tackiness in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters-tackiness, through the subject product perception assessment.
where will you rank the test product in terms of non-sticky/non-oily in which 1 indicate very poor and 5 indicate excellent. | On Day 01 and after test product usage on Day 01 at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameters-non-sticky/non-oily through the subject product perception assessment.
where will you rank the test product in terms of light weight in which 1 indicate very poor and 5 indicate excellent. | On Day 01 after usage of test product at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of change in organoleptic parameter light weight through the subject product perception assessment through the subject product perception assessment.
where will you rank the test product in terms of satisfaction in which 1 indicate very poor and 5 indicate excellent. | On Day 01 after usage of test product at T15 minutes, and on Day 15 (±2 Days)
  To assess the test product in terms of organoleptic parameter in rate in terms of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No